CLINICAL TRIAL: NCT03620110
Title: Prospective Collection of Whole Blood Specimens From Pregnant Women at Any Risk of Fetal Chromosomal Anomaly for the Development of a Noninvasive Prenatal Test
Brief Title: A Study Collecting Blood Samples From Pregnant Women to Aid in the Development of a Noninvasive Prenatal Test
Status: Completed | Type: Observational
Sponsor: Illumina, Inc. (Industry)
Collaborators: Agility Clinical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NIPT-C00-002
Record Dates: First submitted 2018-07-06; First posted 2018-08-08 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human blood specimens will be spun to plasma and stored at -80C freezers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to collect whole blood samples from women with viable pregnancies of at least 10 weeks gestation (at any risk for fetal chromosomal anomaly) for future testing with an investigational noninvasive prenatal test(s) (NIPTs), and to establish clinical truth compared to a clinical reference standard.

DETAILED DESCRIPTION:
This is a prospective, multi-center specimen collection study; each subject's treatment, management, or medical care will not be determined by the study protocol.

Women 18 years of age or older with a viable pregnancy of at least 10 weeks gestation will be enrolled. A whole blood sample will be collected from each subject.

Subjects will be followed until data or specimens used to establish the clinical reference standard are collected, and pregnancy outcome and birth information is collected (if applicable). If cytogenetic test results from standard-of-care procedures are not available and pregnancies end in live births, a neonatal buccal swab specimen will be collected.

Maternal specimens will be processed to plasma and stored for future testing with an investigational NIPT(s). There will be no investigational NIPT results nor centralized CMA LDT results generated under this protocol.

Cytogenetic results from standard-of-care procedures and microarray results will be used to classify the clinical status of subjects according to the clinical reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Has a viable pregnancy of at least 10 weeks, 0 days gestation at the time of maternal specimen collection (singleton or multiple pregnancy acceptable),
* Be 18 years of age or older at enrollment, and
* Is willing and able to provide documentation of informed consent.

Exclusion Criteria:

* Has a prior NIPT result from the current pregnancy,
* Had an invasive prenatal diagnostic procedure (eg, CVS, amniocentesis) in the current pregnancy before maternal specimen collection,
* Has a history of transplant or malignancy,
* Had a transfusion of blood or blood components up to 8 weeks before maternal specimen collection,
* Had preimplantation genetic screening for the current pregnancy (for in vitro fertilization patients only), or
* Has already participated in the study (enrolled previously)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women 18 years of age or older, at any risk of fetal chromosomal anomaly, with a viable pregnancy of at least 10 weeks gestation
Sampling Method: Non-Probability Sample
Enrollment: 2209 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Absence of chromosomal aneuploidy | 12 months
  Collect up to 2,200 maternal blood samples with the number of affected samples with chromosomal aneuploidy less than 0.5% based on clinical data from standard of care invasive procedure, neonate physical exam or chromosomal microarray result from the neonate buccal swab specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Wapner, MD, Principal Investigator — Columbia University
Locations (8):
- United States (8):
  - Valley Perinatal Services, Phoenix, Arizona
  - Unified Women's Clinical Research - Hagerstown, Hagerstown, Maryland
  - United Women's Clinical Research-Greensboro, Greensboro, North Carolina
  - Unified Women's Clinical Research - Morehead City, Morehead City, North Carolina
  - Unified Women's Clinical Research - Raleigh, Raleigh, North Carolina
  - Unified Women's Clinical Research - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Jackson Clinic, Jackson, Tennessee
  - The Group for Women, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No